CLINICAL TRIAL: NCT04848961
Title: Leveraging Mammography to Identify and Engage Women at Risk for Lung Cancer in Lung Cancer Screening
Brief Title: A Study to Develop a Strategy to Increase Lung Cancer Screening in Women Who May Be at Risk for Lung Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-103
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Smoking
Keywords: mammogram; LDCT screening; BiRADS 1; BiRADS 2; 21-103; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women who have had a mammogram (Experimental): Participants will consist of eligible women who have had a mammogram
  Interventions: Behavioral: LungTalk

INTERVENTIONS:
Behavioral: LungTalk — MSK developed LungTalk, a novel computer-tailored health communication and decision support tool to (1) increase awareness and knowledge about lung screening; (2) decrease perceived barriers to screening based upon misinformation; and (3) increase screening rates.

SUMMARY:
The purpose of this study is to develop a digital strategy to increase awareness about lung cancer screening among women who are eligible to receive it. The digital strategy involves email communications and LungTalk, a web-based (accessed through the Internet) health communication tool that uses text, audio, video, and animation to increase awareness and knowledge about lung cancer screening. This study will focus on women who have recently received a screening mammogram.

ELIGIBILITY:
Inclusion Criteria:

* LDCT screening-eligible women who received a BiRADS 1 (negative) or 2 (benign/non-cancerous finding) result from a screening mammogram in the last 7 days
* Age 50-80 years
* ≥ 20-pack-year smoking history of combustible cigarettes as per self report
* Women who currently smoke or quit within past 15 years as per self report
* Lung screening naïve as per self-report

Exclusion Criteria:

* Lung cancer diagnosis
* Chest CT within the last 12 months

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants accrued through digital outreach to identify breast screening participants eligible for lung screening | 6 months
  Develop a proactive digital outreach and engagement strategy to identify breast screening patients who are eligible for lung screening.

CONTACTS AND LOCATIONS:
Overall Officials: Tali Amir, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT04848961/ICF_000.pdf